CLINICAL TRIAL: NCT03550872
Title: Effect of Exercise Training in Patients With Heart Failure and Permanent Atrial Fibrillation
Brief Title: Exercise Training in Patients With Heart Failure and Permanent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Heart of Institute
Record Dates: First submitted 2018-05-23; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: heart failure, atrial fibrillation and exercise training
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: To evaluate the physical effect of physical training in patients with heart failure and permanent atrial fibrillation
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients in the group who are continuously guided as the activities of daily living normally avoiding participation in any regular program of physical exercise does not proceed from the study.
- Training Group (Experimental): the patients randomized to the physical training group will undergo the supervised physical training program
  Interventions: Behavioral: Physical Training

INTERVENTIONS:
Behavioral: Physical Training — Participants will perform physical training three times a week on a stationary bicycle. The exercise intensity will be controlled between 14 and 16 by the Borg Scale for 40 minutes
  Arms: Training Group

SUMMARY:
The positive effect of physical training in patients with heart failure (HF) has been increasingly established. However, the presence of atrial fibrillation (AF), mainly in its permanent form, makes the clinical condition of the patients more compromised.

DETAILED DESCRIPTION:
The positive effect of physical training in patients with heart failure (HF) has been increasingly established. However, the presence of atrial fibrillation (AF), mainly in its permanent form, makes the clinical picture of these patients more compromised. The literature has not yet demonstrated studies involving indication of physical exercise therapy when AF is associated with HF. Thus, the hypothesis is that physical training improves functional capacity, cerebral oxygenation, autonomic aspects, vascular aspects, cardiac function, plasma markers, quality of life and cognitive function of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically stable NYHA class II to III heart failure with permanent atrial fibrillation (AF);
* Left ventricular ejection fraction ≤40%;
* Patients refractory and / or no indication of the treatment of reversal to the rhythm;
* Patients in optimization specific drug therapy for HF and AF.

Exclusion Criteria:

* High-frequency ventricular response;
* Neuromuscular / neuropathy disease;
* Physical and mental impairment;
* Chronic obstructive pulmonary disease;
* Diabetes mellitus;
* Decompensated arterial hypertension;
* Autonomic neuropathy;
* Recent myocardial infarction (<6 months);
* Ventricular arrhythmias;
* Atrial flutter;
* Renal failure;
* Use implantable electronic cardiac device or indication for implantation;
* Pregnancy;
* NYHA Functional Class IV;
* Resting heart rate <55 bpm;
* Wolff Parkinson White Syndrome;
* Thyroid dysfunction;
* Unstable angina;
* Recent history of thromboembolic event;
* Inability to sign the consent form;
* Participation in regular physical training program;
* Use of alcoholic beverages.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06-21; Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Functional Capacity Assessement | two year
  unctional function is assessed by measuring oxygen consumption (VO2). Multidimensional electrocardiography logo will be connected to a computerized system through a remote and tracheal control system. Through Oxygen Detergent (O2) and carbon dioxide (CO2) the concentrations of O2 and CO2, respectively, are analyzed for each respiratory cycle.

SECONDARY OUTCOMES:
Muscle Sympathetic Nervous Activity Assessment | Two year
  Muscle sympathetic nerve activity will be measured by the direct technique of multiple recording units of the efferent postganglionic pathway, the fascicle of the muscular nerve, in the fibular nerve, immediately inferior to the head of the fibula, in the leg. The experiments will be performed in an electrically isolated room with supine individuals. The records will be obtained by implanting a microelectrode on the fibular nerve and a reference microelectrode approximately one to one centimeter away from the first.
Measurement of Muscle Blood Flow | Two year
  The muscular blood flow will be evaluated by the venous occlusion plethysmography technique. The patient will be placed in the dorsal position with the arm elevated above the heart. The silicone-filled mercury-filled tube attached to a low pressure transducer will be placed around the forearm and connected to the plethysmograph.
Evaluation of endothelium-dependent vascular function | Two year
  Endothelium-dependent vascular function will be assessed by muscle vasodilation during isometric manual retention exercise with 30% maximal voluntary contraction for 3 minutes. The level of effort perception will be assessed by the Borg scale.
Evaluation of neurovascular control during mental stress | Two
  After this period, the ANSM, FSM, PA, FC, and FR responses will be evaluated during the application of the Stroop Color Word test. This test consists of a table that has a series of color names, written with an ink different from that of the meaning of the word. The patient should say "high" and as soon as possible in what color the word is written and not the meaning of the word. This procedure will be done as follows: 3 minutes baseline, 4 minutes color test and 2 minutes recovery. At the end of the test will be asked each patient, the degree of difficulty of the color test. This will be done from a standard table of degree of difficulty: 0 = not stressful; 1 = a little stressful; 2 = stressful; 3 = very stressful; 4 = extremely stressful.
Measurement of Pulse Wave Velocity (PWV) | Two year
  VOP will be measured non-invasively using VICORDER® equipment (medical CE, IEC, FDA). Measurements will be obtained using a 100 mm cuff of blood around the thigh to measure the femoral pulse and a partial cuff of 30 millimeters around the neck at the level of the carotid artery. The cuffs will be inflated every 60mmHg, and the high-quality waveforms will be recorded simultaneously for 3 seconds, with the patients positioned in the supine position using a volume-shifting method. The wave impulse transition time will be determined using a cross-correlation algorithm. The length of the path will be defined as the distance between the sternum furcula and the upper part of the thigh sheath as indicated by the manufacturer.
Evaluation of cardiac structure and function | Two year
  For the evaluation of the cardiac function, the patients will be submitted to a one-dimensional (M-mode), two-dimensional transthoracic echocardiographic study with pulsed, continuous and color Doppler echocardiography. The Sequoia 512 (Acuson, Mountain View, CA) will be used with the 2.5-4.0 Mhz 3V2c coupled multifrequency transducer. The exams were recorded on DVD.
  Patients will be positioned and examined. Three electrocardiographic electrodes will be placed on the chest wall for simultaneous recording of the electrocardiogram in the ultrasound system and the parasternal long axis, parasternal short axis, aorta / AE, mitral valve and papillary and apical levels, in 4 and 2 rooms.
Evaluation of the concentration of plasma biomarkers | Two year
  For the determination of the plasma concentration of Norepinephrine (NE), Natriuretic Atrial Peptide (ANP), Cerebral Natriuretic Peptide (BNP), Interleukin-6 (I-6) and Tumor Necrosis Factor- (TNF-alpha) and Angiotensin II, two peripheral blood collections were performed at different times (pre and post training). At each moment 3 ml of blood will be collected in tubes containing EDTA. The supernatant (plasma) will be removed and transferred to two eppendorf microtubes (proof and counter-proof) where they will be stored at -80º C until the moment of analysis. Samples will be quantified at the Genesis Laboratory (São Paulo / SP) using the enzyme immunoassay technique (ELISA) according to standardized laboratory protocols.
Quality of life assessment | Two year
  he Minnesota Living With Heart Failure Questionnaire will be used in its validated Portuguese version74, which evaluates scores of quality of life limitations, addressing the physical, emotional and total score dimensions. It is a questionnaire of 21 questions regarding the limitations that are frequently associated with heart failure and should consider the last month to respond to the questionnaire. The scale of responses for each question ranges from 0 (zero) to 5 (five), where 0 represents without limitations and the maximum limitation. For the physical dimension score is calculated the sum of eight questions (2, 3, 4, 5, 6, 7, 12 and 13) that are highly interrelated with dyspnea and fatigue; the emotional dimension score is composed of five questions (17, 18, 19, 20 and 21); the other questions (1, 8, 9, 10, 11, 14, 15 and 16) added to the questions related to the physical and emotional dimensions, form the total score.
Assessment of cognitive function | Two year
  Cognitive assessment will be performed through the Mini Mental State Examination (MMSE) 75. This questionnaire is used to evaluate the overall cognitive state (general cognitive state) and is divided into seven categories: temporal orientation, spatial orientation, three-word register, attention and calculation, three-word recall, language and visuo-constructive ability. The MMSE has a score of 0 to 30 points, and the lower the score the higher the indication of cognitive decline.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Veiga Guimarães, Principal Investigator — Institute of Heart of the Sao Paulo University
Locations (1):
- Heart Institute of Hospiral Clinics of the University of São Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No